CLINICAL TRIAL: NCT03565952
Title: Effects of Cranial Massage in Menopausal Women With Insomnia
Brief Title: Effects of Cranial Massage in Menopausal Women
Acronym: CM-MWin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID0020
Record Dates: First submitted 2018-05-30; First posted 2018-06-21 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Menopausal Women
Keywords: Menopausal women; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranial massage (Experimental): Manual cranial therapy consisting of massage and cranial relaxing techniques, lasting 30 minutes each session approximately, for 3 weeks and one month follow-up. Manual therapy consists of a prone and supine cranial massage.
  Interventions: Other: Cranial massage
- Control Group (Active Comparator): The control group does not receive treatment.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Cranial massage — Manual cranial therapy consisting of massage and cranial relaxing techniques, lasting 30 minutes each session approximately, for 3 weeks and one month follow-up. Manual therapy consists of a prone and supine cranial massage.
  Arms: Cranial massage
Other: Control group — The control group does not receive treatment
  Arms: Control Group

SUMMARY:
INTRODUCTION Menopause is one more stage in a woman's life. The hormonal change is associated with a series of symptoms that usually manifest around 50 years. Not all women manifest all the symptoms or with the same intensity. The most common symptoms are: hot flushes and night sweats, changes in mood, insomnia or difficulty sleeping, weight gain, vaginal dryness and / or urinary problems; what is detrimental to the well-being of women. At this stage the woman feels more discouraged than usual, and may show moments of anxiety, stress or irritability with the people around her. Sleep disturbances can also cause a state of tiredness and excessive sleepiness during the day, or even persistent headaches that interfere with the daily routine could improve some of these aspects related to sleep disturbances and thus the quality of life of the woman.

The objectives of this study are to know the effect of cranial therapeutic massage on insomnia, in order to improve the quality of life and the woman's corporal satisfaction, and to promote a better functioning and performance of the activities of daily life.

MATERIAL AND METHODS In this study, the investigators selected women aged between 45 and 60 years, who presented changes and symptoms characteristic of the menopausal period, accompanied by alterations in sleep. In addition, the inclusion criteria require that women have not had a menstrual period for one year.

Exclusion criteria are excessive stress, the use of medications to promote sleep and some type of contraindication to receive treatment.

Protocol design It consists of a randomized clinical trial, with a total of 50 participants (n = 50), divided into a control group (n = 25) and an experimental group (n = 25).

Intervention The experimental group is subjected to 1 session per week of manual cranial therapy consisting of massage and cranial relaxing techniques, with a duration of 30 minutes each session approximately, for 3 weeks and one month follow-up. Manual therapy consists of a prone and supine cranial massage.

The control group does not receive treatment, but they will be evaluated the same as the experimental group.

Evaluations Clinical interview Includes anthropometric data (age, weight and height). The quality of life questionnaire Sf-36 and the Menopause Rating Scale (MRS) that assesses the state of well-being of the menopausal woman through 11 simple answer questions.

The Pittsburg Quality of Sleep Questionnaire (PSQI) takes sleep habits into account during the last month. The PSQI contains a total of 19 questions, grouped into 10 questions. In all cases, a score of 0 would indicate ease of sleeping, while a score of 3 would be a severe difficulty.

On the other hand, the Sleep Journal also evaluates sleep habits, characteristics and sleep quality, but unlike the previous one, this questionnaire has to be answered daily by the patients.

The Perceived Stress Scale (PSS) is composed of 14 questions that relate to the level of stress perceived during the last month; The higher the score of each question, the higher the level of stress the person has.

The Body Satisfaction Questionnaire. 10 questions is which must be answered according to the state of health that best describes the person at that time.

The Patient Global Impression of Change Scale questionnaire assesses the sensation of change, in terms of quality of life and sleep, functionality and limitation to perform the activities of daily life, which the participant has experienced since the beginning of the treatment of this study.

Analysis of data The data obtained will be stored in a database (SPSS), with which the analysis of the data will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* women from 45 to 60 years old
* who have not experienced any menstrual cycle for at least one year.
* showing clear menopausal symptoms.

Exclusion Criteria:

* that participants have not used more than twice a week of medication to promote sleep.
* that present contraindications to receive the treatment.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menopausal women with insomnia
Enrollment: 50 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Quality of Sleep | 8 week
  Pittsburg Quality of Sleep Questionnaire (PSQI). The Pittsburg Quality of Sleep Questionnaire (PSQI) takes sleep habits into account during the last month. The PSQI contains a total of 19 questions, grouped into 10 questions. In all cases, a score of 0 would indicate ease of sleeping, while a score of 3 would be a severe difficulty.

SECONDARY OUTCOMES:
Health status | 8 week
  SF-36 is a health questionnaire, both physical and metal. It contains 36 items comprising 8 health status sub-scales. It includes different dimensions (Bodily Pain, Perceptions, Mental Health, Physical Function, Role-physical, Role-emotional, Social Function, and Vitality). Positive and negative health statuses are assessed. To evaluate each dimension, the items are transformed on a scale from 0 to 100. The result is obtained by summation of all the questions, in which 0 is the worst and 100 the best result and state of health.
Climacteric symptoms | 8 week
  The Menopause Rating Scale (MRS) assesses the severity of climacteric symptoms. It consists of 11 symptoms divided into three groups: 1. MRS somatic level, includes: hot flashes, sweating, heart discomfort, sleep disturbances and joint and muscle discomfort; 2. Psychological MRS: depressive mood, irritability, anxiety and physical and mental fatigue; 3. Urogenital MRS: sexual problems, problems with urine and vaginal dryness.
  It is an easy-to-complete questionnaire, in which each participant must attribute to each clinical manifestation a score of 0 to 4, depending on whether he or she experiences the described symptoms with greater or lesser intensity. The total MRS score is the sum of the scores obtained in each block.
Body Satisfaction | 8 week
  Body Satisfaction and global self-perception Questionnaire. It contains 10 positive and 10 negative adjectives about the participant's body sensation with alternative answers ranging from 1 = Excellent to 5 = Poor. Each question is scored independently.
Perceived Stress | 8 week
  Perceived Stress Scale (PSS). It consists of 14 questions that relate to the level of perceived stress during the last month. Each item has a score of 0 to 4 (0 = never, 1 = almost never, 2 = occasionally, 3 = often, 4 = very often). The total PSS score is the sum of the results of each item, which indicates that the higher the score attributed to each question, the higher the level of stress that the person presents.
Global Impression of Change | 8 week
  Patient Global Impression of Change Scale, published by Hurst H. and Bolton J. Evaluates the sensation of change after the treatment received. It contains 7 affirmations (1 = I have improved a lot, 2 = I have improved a lot, 3 = I have improved a little, 4 = I am the same, 5 = I have worsened a little, 6 = I have worsened a lot, 7 = I have worsened a lot), together with an analog scale on the degree of change (0 = much better, 5 = no change, 10 = much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Valencia, Spain